CLINICAL TRIAL: NCT01024270
Title: Cervical Priming With Misoprostol Prior to Operative Hysteroscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Duk Soo Bae/Chairman of Dept. of Ob. & Gyn, Samsung Medical Center
Allocation: Randomized | Masking: Single
Other Study IDs: 2008-06-035
Record Dates: First submitted 2009-11-12; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-07

CONDITIONS: Cervical Ripening
Keywords: endometrial pathology of uterus; operative hysteroscopy; efficacy of misoprostol per different routes
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Care Provider

ARMS (1):
- sublingual, oral and vaginal administration of misoprostol (Experimental)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol

SUMMARY:
The primary outcome measure in this study was the preoperative cervical width after misoprostol administration. The secondary outcomes were duration of cervical dilatation, up to Hegar number 10, complications during cervical dilation and the hysteroscopy, and misoprostol associated side effects. The cervical width was assessed by performing cervical dilatation, starting with a number 10 Hegar dilator and subsequently inserting smaller Hegar dilatators until the dilator could pass through the internal os without resistance. The largest one that could be passed was recorded as the initial cervical width.

The mean cervical diameter, after oral and vaginal misoprostol of 400 μg, has been reported to be 6.0 ± 1.5 mm and 7.3 ± 1.6 mm, respectively 4. The investigators hypothesized that equivalence was of clinical significance if the difference in the initial cervical width was less than 1 mm among groups with the standard deviation of the initial cervical width of 1.6 mm. The estimated sample size was 47 patients in each group; this would be able to detect an equivalent effect in the groups with a power of 80% and a type 1 error (a) of 0.017. Data are expressed as the mean ± SD (standard deviation) or median with range or as the number (%) of cases.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients that were suspected as having intrauterine pathology such as submucosal myoma, endometrial polyps or other endometrial pathological findings based on the transvaginal ultrasound were enrolled.
* women who are more than 20 years of age with having sexual contact history
* women whose last menstrual period are within the last two months.

Exclusion Criteria:

* Post menopausal women
* any evidence of a contraindication or allergy to PGs
* any sign of genital infection, history of cervical surgery, endometrial lesions with suspected endo- or exocervical lesions that could affect the cervical resistance or patients that were not candidates for surgery.

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure in this study was the preoperative cervical width after misoprostol administration. | 1 year

SECONDARY OUTCOMES:
Duration of cervical dilatation, up to Hegar number 10. | 1 year
Complications during cervical dilation. | 1 year
Misoprostol associated side effects. | 1 year
Complications during the hysteroscopy. | 1

CONTACTS AND LOCATIONS:
Overall Officials: Duk Soo Bae, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee YY, Kim TJ, Kang H, Choi CH, Lee JW, Kim BG, Bae DS. The use of misoprostol before hysteroscopic surgery in non-pregnant premenopausal women: a randomized comparison of sublingual, oral and vaginal administrations. Hum Reprod. 2010 Aug;25(8):1942-8. doi: 10.1093/humrep/deq083. Epub 2010 Jun 11. PMID 20542898